CLINICAL TRIAL: NCT02604550
Title: Comparison Between Femoral Nerve Block and Adductor Canal Block for Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Controlled Trial
Brief Title: Anterior Cruciate Ligament Pain Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Xerogeanes, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00083740
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — oxycodone-acetaminophen; Naproxen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): Subjects undergoing anterior cruciate ligament (ACL) surgery will be randomized to receive 20 mL of ropivacaine 0.5% in the femoral nerve. Subjects will also receive standard of care Percocet 7.5/325 and naprosyn following surgery.
  Interventions: Drug: Ropivacaine 0.5%; Drug: Percocet 7.5/325; Drug: Naprosyn 500 mg
- Adductor Canal Block (Active Comparator): Subjects undergoing anterior cruciate ligament surgery will be randomized to receive 20 mL of ropivacaine 0.5% in the adductor canal. Subjects will also receive standard of care Percocet 7.5/325 and naprosyn following surgery.
  Interventions: Drug: Ropivacaine 0.5%; Drug: Percocet 7.5/325; Drug: Naprosyn 500 mg

INTERVENTIONS:
Drug: Ropivacaine 0.5% — Ropivacaine 0.5% will be administered to the femoral nerve or adductor canal.
Drug: Percocet 7.5/325 — Percocet 7.5/325 will taken as needed up to every four hours.
Drug: Naprosyn 500 mg — Naprosyn 500 mg will be taken twice daily.

SUMMARY:
The objective of this study is to compare the pain control benefit of two different types of nerve blocks in patients undergoing anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, surgeon-blinded, two-armed trial to investigate the safety and efficacy of femoral nerve blocks versus adductor canal blocks for participants undergoing outpatient anterior cruciate ligament (ACL) reconstruction surgery.

The objective of this study is to compare the pain control benefit of two different types of nerve blocks. Ropivacaine, which is FDA-approved for use in both femoral nerve blocks as well as adductor canal blocks, will be utilized. The study will be comparing the efficacy between FDA approved treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled anterior cruciate ligament (ACL) surgery at the Emory Orthopaedic and Spine Center
* Patients willing and able to provide written informed consent
* Parents willing and able to provide written informed consent for minors

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with liver dysfunction or renal failure
* Patients with a known allergy to ropivacaine
* Patients with a local infection
* Patients who take chronic pain medications
* Patients with an opioid tolerance
* Patients with known coagulopathy or bleeding risk.
* Patients who are getting neuraxial anesthesia for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Xerogeanes, MD, Principal Investigator — Emory University
Locations (1):
- Emory Healthcare Orthopaedics and Spine Center, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing scheduled anterior cruciate ligament (ACL) surgery at the Emory Orthopaedic and Spine Center in Atlanta, Georgia were prospectively randomized to receive either a femoral nerve block (FNB) or an adductor canal block (ACB). Participants were enrolled between December 2015 and April 2016.
Groups:
- Femoral Nerve Block: Participants randomized to receive 20 milliliter (mL) of ropivacaine 0.5% in the femoral nerve.
- Adductor Canal Block: Participants randomized to receive 20 milliliter (mL) of ropivacaine 0.5% in the adductor canal
Period: Overall Study
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Started | 56 | 59
Completed | 31 | 33
Not Completed | 25 | 26
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incomplete data using paper journal | 18 | 19

BASELINE CHARACTERISTICS:
Population: All participants who consented to take part in the trial and received the intervention of the study arm they were randomized to.
Groups:
- Femoral Nerve Block: Participants randomized to receive 20mL of ropivacaine 0.5% in the femoral nerve.
- Adductor Canal Block: Participants randomized to receive 20mL of ropivacaine 0.5% in the adductor canal
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block | Adductor Canal Block | Total
Number analyzed (Participants) | 56 | 59 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 17 | 31
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 25 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 35 | 78
  Unknown or Not Reported | 13 | 24 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 13 | 28
  White | 26 | 21 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 24 | 37
Region of Enrollment [Number; unit: participants]
  United States | 56 | 59 | 115

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain scores range from 0 (no pain at all) to 10 (worst imaginable pain). Pain level was reported at the time of discharge from the surgery recovery room, the evening of the day of surgery, and then three times per day for six days post-surgery. During the six days after surgery, the morning assessment asked about typical knee pain levels overnight, the afternoon assessment asked about knee pain levels since the morning entry, and the evening assessment asked about knee pain levels since the afternoon entry.
Time Frame: Post-surgery (day of surgery to 6 days post-surgery)
Population: This analysis includes participants who completed the study and used a smartphone application to record pain level for 6 days post-surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
units on a scale
  Recovery room discharge | 4.1 (1.8) | 4.0 (2.8)
  Day of surgery, evening | 3.9 (2.2) | 5.1 (2.9)
  Post-surgery Day 1 - Morning | 5.7 (2.6) | 5.7 (2.4)
  Post-surgery Day 1 - Afternoon | 5.1 (2.3) | 5.0 (1.8)
  Post-surgery Day 1 - Evening | 5.5 (2.3) | 6.0 (2.1)
  Post-surgery Day 2 - Morning | 5.4 (2.3) | 5.3 (2.3)
  Post-surgery Day 2 - Afternoon | 4.5 (1.9) | 4.6 (1.8)
  Post-surgery Day 2 - Evening | 4.3 (2.0) | 4.5 (2.1)
  Post-surgery Day 3 - Morning | 4.2 (2.0) | 4.0 (3.1)
  Post-surgery Day 3 - Afternoon | 3.8 (1.9) | 3.4 (2.5)
  Post-surgery Day 3 - Evening | 4.0 (2.1) | 3.7 (2.3)
  Post-surgery Day 4 - Morning | 3.5 (2.2) | 3.0 (2.2)
  Post-surgery Day 4 - Afternoon | 3.2 (2.1) | 2.7 (2.0)
  Post-surgery Day 4 - Evening | 4.0 (2.4) | 3.3 (2.4)
  Post-surgery Day 5 - Morning | 3.7 (2.2) | 3.1 (2.1)
  Post-surgery Day 5 - Afternoon | 3.6 (2.1) | 3.3 (2.2)
  Post-surgery Day 5 - Evening | 3.4 (2.3) | 3.3 (2.4)
  Post-surgery Day 6 - Morning | 3.7 (2.2) | 3.1 (2.2)
  Post-surgery Day 6 - Afternoon | 3.2 (1.6) | 3.2 (2.0)
  Post-surgery Day 6 - Evening | 2.7 (1.6) | 2.8 (2.2)

2. Secondary Outcome: Number of Percocet Tablets Consumed
Description: Participants recorded the total number of Percocet 7.5/325 (acetaminophen and oxycodone) tablets they took every day, in order to assess post-surgical use of opioids between the study arms,
Time Frame: Post surgery, Day 0 to Day 6
Population: This analysis includes participants who completed the study and used a smartphone application to record the number of Percocet tablets taken for 6 days post-surgery.
Measure: Mean (Standard Deviation); unit: count of tablets
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
count of tablets
  Day of surgery (Day 0) | 2.0 (1.2) | 2.4 (1.7)
  Post-surgery Day 1 | 4.6 (2.5) | 4.7 (2.9)
  Post-surgery Day 2 | 3.7 (2.6) | 3.6 (2.6)
  Post-surgery Day 3 | 2.3 (1.9) | 2.2 (2.2)
  Post-surgery Day 4 | 1.1 (1.3) | 1.2 (2.1)
  Post-surgery Day 5 | 0.6 (1.4) | 1.4 (1.5)
  Post-surgery Day 6 | 0.3 (0.7) | 0.4 (0.7)

3. Secondary Outcome: Total Hours of Sleep
Description: The total hours of sleep first postoperative night, between 0 to 12 hours.
Time Frame: First Postoperative Night (up to 12 hours)
Population: This analysis includes participants who completed the study and used a smartphone application to record their number of hours of sleep during the night following their surgery.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
hours | 6.3 (2.0) | 5.8 (1.4)

4. Secondary Outcome: Patient-Reported Nausea
Description: Total occurrences of patient-reported nausea post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants completing the study who used a smartphone application for 6 days post-operatively to record every time they experienced nausea.
Measure: Number; unit: occurrence of nausea
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
occurrence of nausea | 3 | 2

5. Secondary Outcome: Patient-Reported Vomiting
Description: Total occurrences of patient-reported vomiting post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants who completed the study and used a smartphone application for 6 days post-operatively to record every time they experienced vomiting.
Measure: Number; unit: occurrence of vomiting
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
occurrence of vomiting | 1 | 1

6. Secondary Outcome: Patient-Reported Constipation
Description: Total occurrences of patient-reported constipation post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants completing the study and who used a smartphone application for 6 days post-operatively to record every time they experienced constipation.
Measure: Number; unit: occurrence of constipation
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
occurrence of constipation | 2 | 1

7. Secondary Outcome: Patient-Reported Sedation
Description: Total occurrences of patient-reported feelings of sedation post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants who completed the study and used a smartphone application for 6 days post-operatively to record every time they experienced feelings of sedation.
Measure: Number; unit: occurrence of sedation
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
occurrence of sedation | 0 | 0

8. Secondary Outcome: Patient-Reported Itching
Description: Total occurrences of patient-reported itching post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants who completed the study and used a smartphone application for 6 days post-operatively to record every time they experienced itching.
Measure: Number; unit: occurrence of itching
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
occurrence of itching | 2 | 1

9. Secondary Outcome: Time to Straight Less Raise
Description: The amount of time (in hours) it takes for participants to have the ability to perform a straight leg raise post-surgery.
Time Frame: Post-Surgery (up to 6 days)
Population: This analysis includes participants who completed the study and used a smartphone application to record when they were able to perform a straight leg raise following surgery.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
hours | 31.7 (26.1) | 16.4 (10.5)

10. Secondary Outcome: Percent of Patients Rating Their Satisfaction as "Excellent" or "Good"
Description: Patient satisfaction will be reported on a scale of excellent, good, satisfactory, or poor, two weeks following surgery.
Time Frame: 2 Weeks Post-Surgery
Population: This analysis includes participants who completed the study and used a smartphone application to record study outcome measures following surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Femoral Nerve Block | Adductor Canal Block
Number analyzed (Participants) | 31 | 33
percentage of participants | 39 | 64

ADVERSE EVENTS:
Time Frame: Data regarding adverse events were collected from the time a participant gave informed consent to take part in the study until the end of the study follow up.
Description: Any change from baseline considered by the investigator to be an untoward medical occurrence different from the standard of care, was reported as an adverse event. Any change from baseline considered by the investigator to be part of the normal daily fluctuations of the underlying disease process, was not reported as an adverse event.
Arm/Group | Femoral Nerve Block | Adductor Canal Block
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/59
Other Adverse Events (participants affected / at risk) | 0/56 | 0/59

LIMITATIONS AND CAVEATS:
Data collection with a paper journal was low, resulting in the study switching to a smartphone application for participant record keeping. The data analyses include participants who enrolled after the smartphone application became available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes